CLINICAL TRIAL: NCT07022171
Title: Physiological and Molecular Mechanisms of Transcutaneous Auricular Vagus Nerve Stimulation in Depression
Brief Title: Mechanisms of Transcutaneous Auricular Vagus Nerve Stimulation in Depression
Acronym: AddVNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 24-0985
Record Dates: First submitted 2025-05-09; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder; Bipolar Disorder
Keywords: transcutaneous; auricular; vagus nerve stimulation; biomarkers; depression
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder; Depression

STUDY DESIGN:
Intervention Model Description: Patients from the clinic of Max-Planck-Institute of Psychiatry are block wise randomly assigned to one of 2 study arms (transcutaneous auricular vagus nerve stimulation, sham transcutaneous auricular vagus nerve stimulation) after they have given informed consent
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tVNS-arm (transcutaneous auricular vagus nerve stimulation) (Experimental): Half of the patients are randomized to the arm receiving transcutaneous auricular vagus nerve stimulation in addition to their regular treatment for a period of six weeks
  Interventions: Device: transcutaneous auricular vagus nerve stimulation
- sham tVNS-arm (sham transcutaneous auricular vagus nerve stimulation) (Sham Comparator): Half of the patients are randomized to the arm receiving sham transcutaneous auricular vagus nerve stimulation in addition to their regular treatment for a period of six weeks. The procedures for sham tVNS will be identical to tVNS, with the only exception that the sham tVNS will be performed with no current output
  Interventions: Device: sham transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation — Half of the patients are randomized to the arm receiving transcutaneous auricular vagus nerve stimulation for a period of six weeks. Transcutaneous auricular vagus nerve stimulation will be carried out as an adjuvant, i.e. in addition to the regular treatment of the participants. The intervention will take place three times a day from Monday to Friday. Each of the three daily sessions is going to last 30-60 minutes, depending on patient tolerance.
  Arms: tVNS-arm (transcutaneous auricular vagus nerve stimulation)
Device: sham transcutaneous auricular vagus nerve stimulation — Half of the patients are randomized to the arm receiving sham transcutaneous auricular vagus nerve stimulation for a period of six weeks. Sham transcutaneous auricular vagus nerve stimulation will be carried out as an adjuvant, i.e. in addition to the regular treatment of the participants. The intervention will take place three times a day from Monday to Friday. Each of the three daily sessions is going to last 30-60 minutes. The procedures for sham tVNS will be identical to tVNS, with the only exception that the sham tVNS will be performed with no current output
  Arms: sham tVNS-arm (sham transcutaneous auricular vagus nerve stimulation)

SUMMARY:
Invasive vagus nerve stimulation (VNS) is an approved treatment of treatment-resistant depression (TRD) in Europe and in USA. Because of the associated possible surgical complications as well as side effects, invasive VNS is applied limitedly in the treatment of depression. Transcutaneous auricular VNS (tVNS), on the other hand, is a non-invasive alternative to traditional invasive VNS. tVNS is still considered an experimental treatment for depression. This is due to the limited high-quality evidence from randomized clinical studies, the not yet fully understood biological mechanisms of action, along with overall limited knowledge about the optimal stimulation parameters. To address these issues, the AddVNS study was initiated. The AddVNS study intends to recruit n=86 patients of the Max Planck Institute of Psychiatry with depression. The patients participating in the AddVNS study are going to receive either tVNS or sham tVNS for a period of 6 weeks. The primary objective of the study is to identify biological, psychological, socio-economic, and clinical biomarkers associated with treatment progression and response to treatment in patients with depression undergoing tVNS. To achieve this, an exploratory design with an assessment of many different parameters including psychophysiology, imaging, blood-based multi-omics, microbiome, psychometrics and neuropsychology will be used.

DETAILED DESCRIPTION:
Background:

Depression is one of the most prevalent mental disorders worldwide and is associated with the highest burden of disease among all psychiatric disorders. Invasive vagus nerve stimulation (VNS) has been approved for the treatment of treatment-resistant depression (TRD). However, invasive VNS is applied limitedly in the treatment of depression due to the associated possible surgical complications and side effects. Transcutaneous auricular VNS (tVNS), on the other hand, is a non-invasive alternative to invasive VNS. During the last decade, the effects of tVNS have been examined in an increasing number of clinical trials across many different disorders, with depression being one of the most prominent areas of interest. Nevertheless, tVNS is still considered an experimental treatment for depression. Reasons for this categorization come from the limited high-quality evidence from randomized clinical studies, the not yet fully understood biological mechanisms of action, along with overall limited knowledge about the optimal stimulation parameters. To address these issues, we initiated the AddVNS study. The primary objective of the study is to identify biomarkers of tVNS and to better understand its biological mechanisms of action in the treatment of depression.

Material and methods:

The AddVNS is a monocentric, exploratory-prospective, randomized, double-blind, sham-controlled interventional study that recruits adult and legally competent patients with current MDD or bipolar disorder with current depression who are treated in MPIP (either inpatient or day clinic treatment). The participants are going to receive either tVNS or sham tVNS for a period of 6 weeks. Both tVNS and sham tVNS will be carried out as an adjuvant, i.e. in addition to the regular treatment of the participants. The intervention will take place three times a day from Monday to Friday. Each of the three daily sessions is going to last 30-60 minutes, depending on patient tolerance. The procedures for sham tVNS will be identical to tVNS, with the only exception that the sham tVNS will be performed with no current output. Participants and investigators are blinded to the assignment of participants to a study arm, except for the investigators responsible for the stimulation. The AddVNS study includes a wide range of assessments, which will be identical for both study arms. Psychophysiological measurements (pupillometry, respiratory rate, 3-channel ECG, skin conductance level, photoplethysmography and an electrogastrogram) will be conducted at baseline, after 3 weeks of intervention and at the end of the 6-week intervention (for a small number of patients, two additional psychophysiological measurements are planed). Actigraphy will take place throughout the 6-week intervention. Two MRI scans are planned over the course of the AddVNS study; one scan is scheduled at baseline and one after the 6-week intervention. Participants will have a total of three venous blood samples taken over the course of the 6-week intervention. They will be asked to collect stool samples that will be used for microbiome analysis at baseline, after 3 weeks of intervention and at the end of the 6-week intervention. Participants will be also asked to fill out self-rating questionnaires (patient health questionnaire 9 and 15, Beck Depression Inventory II, Snaith-Hamilton-Pleasure-Scale, Questionnaire for complaints of cognitive disturbances) once a week, while two further questionnaires will be obtained at baseline and after the 6-week intervention (Rejection Sensitivity Questionnaire, World Health Organization Disability Assessment Schedule questionnaire). During a clinical interview at baseline, after 3 weeks of intervention and after 6 weeks of intervention, clinician-rating scales (Montgomery-Åsberg Depression Rating Scale, Hamilton Rating Scale for Depression with 21 items, Hamilton Rating Scale for Anxiety, Global Assessment of Functioning) will be obtained. Furthermore, a neuropsychological assessment is carried out at baseline and after the 6-week intervention, while a personality assessment will be performed at baseline. To assess the longitudinal effects of tVNS, we will ask the patients to fill out self-rating questionnaires (patient health questionnaire 9 and 15, Beck Depression Inventory II, Snaith-Hamilton-Pleasure-Scale, Questionnaire for complaints of cognitive disturbances, Rejection Sensitivity Questionnaire, World Health Organization Disability Assessment Schedule questionnaire) 6 and 12 weeks after the end of the intervention.

Discussion:

Taken together, the main goal of the AddVNS study is to identify biological, psychological, socio-economic, and clinical biomarkers associated with treatment progression and response to treatment in patients with depression undergoing tVNS. The strength of the study lies in its study design, as AddVNS is a randomized controlled trial combining a meticulous documentation of the tVNS procedure with a wide assessment of many different parameters. This makes the AddVNS study one of the most extensive studies of tVNS in depression to date.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65 years, legally competent and able to provide informed consent;
2. diagnosis of a depressive episode (MDD or bipolar disorder) according to DSM 4/DSM 5 or ICD-10/ICD-11;
3. signed informed consent documents for the AddVNS study;
4. signed informed consent and participation in the biobanking project of MPIP;
5. use of a safe contraceptive method

Exclusion Criteria:

1. age < 18 years or age > 65 years;
2. pregnancy or planning to get pregnant during the study period, breastfeeding;
3. legal supervision;
4. pervasive developmental disorders and/or intellectual disability;
5. acute substance abuse (e.g., alcohol, prescription or illicit drugs);
6. severe neurological disease;
7. technically or anatomically not possible tVNS (e.g., microtia or anotia, vagotomy);
8. current treatment with an established neurostimulation method (e.g., ECT, rTMS, VNS);
9. metallic foreign bodies, implanted intracranial devices or cerebral shunts;
10. severe general illness (e.g., relevant anemia requiring transfusion, high-grade cardiac arrythmia, severe cardiomyopathy);
11. active implants (e.g., cochlear implant, cardiac pacemaker, implantable cardioverter-defibrillator)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2030-03-17 (Estimated); Study Completion 2030-03-17 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pupillometry | Baseline, week 3, week 6
  Pupil diameter associated with the clinical response to tVNS
Change from baseline in 3-channel ECG | Baseline, week 3, week 6
  3-channel ECG associated with the clinical response to tVNS
Change from baseline in skin conductance level | Baseline, week 3, week 6
  Skin conductance level associated with the clinical response to tVNS
Change from baseline in photoplethysmography | Baseline, week 3, week 6
  Photoplethysmography associated with the clinical response to tVNS
Change from baseline in electrogastrogram | Baseline, week 3, week 6
  Electrogastrogram associated with the clinical response to tVNS
Change from baseline in the functional status of brainstem nuclei | Baseline, week 6
  Functional status of selected brainstem nuclei (by fMRI) associated with the clinical response to tVNS
Change from baseline in the response patterns in the reward anticipation task | Baseline, week 6
  Response patterns in the reward anticipation task (by fMRI) with the clinical response to tVNS
Change from baseline in motor activity | Continuously starting from baseline up to week 6
  Motor activity changes, measured by actigraph, associated with the clinical response to tVNS
Change from baseline in heart rate | Continuously starting from baseline up to week 6
  Heart rate, measured by actigraph, associated with the clinical response to tVNS
Change from baseline in heart rate variability | Continuously starting from baseline up to week 6
  Heart rate variability, measured by actigraph, associated with the clinical response to tVNS
Change from baseline in oxygen saturation | Continuously starting from baseline up to week 6
  Oxygen saturation, measured by actigraph, associated with the clinical response to tVNS
Change from baseline in skin temperature | Continuously starting from baseline up to week 6
  Skin temperature, measured by actigraph, associated with the clinical response to tVNS
Investigation of gene expression changes | Baseline, week 3, week 6
  Gene expression changes over time (based on material extracted from peripheral blood)
Investigation of epigenetic changes | Baseline, week 3, week 6
  Epigenetic changes over time (based on material extracted from peripheral blood)
Investigation of protein changes | Baseline, week 3, week 6
  Protein changes over time (based on material extracted from peripheral blood)
Investigation of lipid changes | Baseline, week 3, week 6
  Lipid changes over time (based on material extracted from peripheral blood)
Investigation of electrolyte changes | Baseline, week 3, week 6
  Electrolyte changes over time (based on material extracted from peripheral blood)
Investigation of immunophenotypic changes | Baseline, week 3, week 6
  Immunophenotypic changes over time (based on material extracted from peripheral blood)
Microbiome changes | Baseline, week 3, week 6
  Microbiome changes (bacteria strains and metabolites) over time
Genetics | Baseline
  Genotyping based on material extracted from peripheral blood

SECONDARY OUTCOMES:
Change from baseline in the Hamilton Depression Rating Scale (HAM-D) | Baseline, week 3, week 6
  The HAM-D measures the presence and severity of depression. Each of the items is rated by a study clinician or trained study staff member and added up to a summary score. Treatment response is generally defined by 50% score reduction, while remission is commonly assumed if the HAM-D score is ≤ 7 points
Change from baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline, week 3, week 6
  The MADRS measures the presence and severity of depression. Each of the terms is rated by a study clinician or trained study staff member and added up to a summary score. Treatment response is generally defined by 50% score reduction, while remission is commonly assumed if the MADRS score falls short of 12 points
Change from baseline in the Global Assessment of Functioning (GAF) | Baseline, week 3, week 6
  The GAF approximates the level of symptom burden and psychosocial as well as occupational functioning in daily life. It is tailored primarily to psychiatric patients. It is rated from 0 to 100 by a trained clinician. The GAF score is a continuous variable and allows to estimate symptom reduction and functional assessment from a foreign rater perspective
Change from baseline in the Beck-Depression-Inventory II (BDI-II) | Weekly up to week 6, week 12, week 18
  The BDI-II measures the presence and severity of depression symptoms on a mostly psychological and partially somatic level. Each of the 21 items is rated by the patient and added up to a summary score. Treatment response is generally defined by 50% score reduction, while remission is commonly assumed if the BDI-II score is ≤ 10 points
Change from baseline in the Patient Health Questionnaire 9 (PHQ-9) | Weekly up to week 6, week 12, week 18
  The PHQ-9 is a brief measure of depression symptoms. Each of the 9 items is rated by the patient from 0 = not at all to 3 = nearly every day and added up to a summary score. Treatment response is generally defined by 50% score reduction, while remission is commonly assumed if the PHQ-9 score is ≤ 5 points.
Change from baseline in the Patient Health Questionnaire 15 (PHQ-15) | Weekly up to week 6, week 12, week 18
  The PHQ-15 is a measure of somatic symptom load in psychiatric disorders. Each of the 15 somatic symptoms is rated by the patient from 0 = not affected to 2 = strongly affected and added up to a summary score. Cut-off values are ≥ 5points (mild), ≥ 10 points (moderate), ≥ 15 points (severe) and represent somatization.
Change from baseline in the Questionnaire on Mental Capacity (FLEI = Questionnaire for Complaints of Cognitive Disturbances ) | Weekly up to week 6, week 12, week 18
  The FLEI measures neurocognitive functioning in the following domains: attention, memory, executive function, control scale. Each of the 35 questions is answered by the patient from 0 = never to 4 = very often. Summary scores are computed for the different neurocognitive domains. Since the FLEI is primarily a continuous variable, symptom reduction is commonly assessed quantitatively
Change from baseline in the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0.) questionnaire | Baseline, week 6, week 12, week 18
  The WHODAS 2.0. questionnaire is a self-rating instrument with 36 items for the assessment of health, functioning, disability and health-related quality of life which can be used across all diseases
Change from baseline in the Rejection Sensitivity Questionnaire (RSQ) | Baseline, week 6, week 12, week 18
  The German modified version of RSQ with 20 items will be used as a measure of rejection sensitivity (RS) to explore the role of RS in the context of tVNS in depressive disorders.
Change from baseline in Snaith-Hamilton-Pleasure-Scale (SHAPS-D) | Weekly up to week 6, week 12, week 18
  SHAPS-D is an instrument for the assessment of anhedonia. Each of the 14 items is rated by the patient and added up to a summary score. Anhedonia is commonly assumed if the SHAPS-D score is > 2.
Change from baseline in Hamilton Rating Scale for Anixety (HAM-A) | Baseline, week 3, week 6
  HAM-A is a rating scale for the assessment of anxiety symptoms. Each of the 14 items is rated by a study clinician or trained study staff and added up to a summary score with a total range from 0 to 56. Remission of anxiety is commonly assumed if the HAM-A score is ≤ 7.
Change from baseline in Trail Making Test Version A (TMT-A) and B (TMT-B) | Baseline, week 6
  TMT is an attention test from COGBAT basic cognitive testing. In the A version, the patient is given the task of connecting circles with the numbers 1 to 25 as quickly as possible in ascending order. This is followed by the B version of the test, in which the patient has to connect circles with the numbers from 1 to 13 and letters from A to L alternatingly in ascending order.
Change from baseline in TOL-F test (Tower of London - Freiburg version) | Baseline, week 6
  TOL-F is a test for planning ability from COGBAT basic cognitive testing. In this task, the patient must move balls on wooden sticks in the fewest number of moves possible so that the specified target condition is reached.
Change from baseline in Episodic memory test | Baseline, week 6
  A short text is read aloud and the patient is asked to memorize the content. The patient is asked to repeat the text immediately after it has been read aloud and again after 30 minutes.
Change from baseline in the INHIB test (Response inhibition) | Baseline, week 6
  INHIB is a test for response inhibition from the COGBAT basic cognitive testing. In this task, circles and triangles are preset. Whenever the triangle appears, the patient must press a button as quickly as possible (go trial), ignoring the circles (no-go trial).
Change from baseline in N-back-verbal test (NBV) | Baseline, week 6
  N-back is a test for working memory from COGBAT basic cognitive testing. The patient is presented with a sequence of letters on a screen and should press a button when the presented letter is the same as the letter before.
Change from baseline in WAF test (perception and attention functions battery ) | Baseline, week 6
  WAF is a test baterry for the assessment of sub-functions of attention and is part of the COGBAT basic cognitive testing. In the AddVNS study the test for cross-modal visual /auditory attention and the test for intrinsic (visual) alertness are used. In the task for cross-modal visual/auditory attention, the patient concentrates simultaneously on a figure and on an auditory stimulus. The intensity of the stimuli changes at certain intervals. The patient must react as soon as one of the two stimuli becomes brighter or quieter twice in a row. In the task for intrinsic (visual) alertness, the patient has to press a button as quickly as possible as soon as a black circle appears on the screen.
Change from baseline in MWT-B test (multiple-choice vocabulary intelligence test B ) | Baseline, week 6
  MWT-B is a multiple choice vocabulary intelligence test. In this test, the patient is given 37 rows with five words each, only one of which actually exists and should be crossed out accordingly.

OTHER OUTCOMES:
Identification of clinical predictors of treatment response namely maladaptive personality traits measured by the German version of the Personality Inventory for DSM-5 and ICD-11 - brief form -version 1.1 (self-rating) | Baseline
  Lead to identification of maladaptive personality traits, no score on a scale.
Identification of clinical predictors of treatment response namely maladaptive personality traits measured by the Levels of Personality Functioning Scale-Brief Form 2.0 (self-rating) | Baseline
  Lead to identification of maladaptive personality traits, no score on a scale.
Sociodemographic variables (age, gender, marital status, income, education, occupation, family history of migration) | Baseline
  Sociodemographic variables as covariables for analysis of treatment response
Medical history (psychiatric history, somatic medical history, family history, substance use history, medication history) | Baseline
  Medical history as covariable for analysis of treatment response
Actual medication | weekly up to week 6
  Reporting of actual medication as covariable for analysis of treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Peter Falkai, MD, Principal Investigator — Max-Planck-Institute of Psychiatry
Locations (1):
- Max Planck Institute of Psychiatry, Munich, Germany